CLINICAL TRIAL: NCT02894840
Title: A Phase I/II Randomized Double Blind Controlled Study to Evaluate the Safety and Immunogenicity of GPO Seasonal Trivalent Inactivated Split Virion Influenza Vaccine in Healthy Thai Adults Aged Between 18 Years to 49 Years
Brief Title: Safety and Immunogenicity of GPO Seasonal Trivalent Inactivated Influenza Vaccine in Healthy Thai Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: The Government Pharmaceutical Organization (Other Government); World Health Organization (Other)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Prof., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GPO Tri Fluvac Vaccine
Record Dates: First submitted 2016-08-24; First posted 2016-09-09 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Influenza
Keywords: GPO Tri Fluvac Vaccine; Tri Fluvac Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- an inactivated influenza vaccine (Active Comparator): 20 volunteers in phase I study and 200 volunteers in phase II study will receive a single dose of a seasonal trivalent inactivated split virion influenza vaccine [A/California/7/2009, reassortant virus NYMC X-181 (H1N1), A/Victoria/210/2009, reassortant virus NYMC X-187 (H3N2), and B/Brisbane/60/2008, reassortant virus NYMC BX-35 virus strains] will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm.
  Interventions: Biological: an inactivated influenza vaccine
- Placebo (Placebo Comparator): 20 volunteers in phase I study and 100 volunteers in phase II study will receive a single dose of placebo will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: an inactivated influenza vaccine — The vaccine will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm.
  Arms: an inactivated influenza vaccine
Other: Placebo — The placebo will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm.
  Arms: Placebo

SUMMARY:
The study is aim to evaluate the safety and immunogenicity of one dose (15 μg HA per strain per dose) of the GPO seasonal trivalent inactivated split virion influenza vaccine (Tri Fluvac) in healthy adults aged 18 to 49 years over 90 days post-injection.

DETAILED DESCRIPTION:
This is a double blind randomized study consisting of two phases - Phase I and Phase II. The same vaccine, a seasonal trivalent inactivated split virion influenza vaccine [A/California/7/2009, reassortant virus NYMC X-181 (H1N1), A/Victoria/210/2009, reassortant virus NYMC X-187 (H3N2), and B/Brisbane/60/2008, reassortant virus NYMC BX-35 virus strains] will be given in both Phase I and Phase II of the study.

The vaccine will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm. After vaccination volunteers will remain at the clinic for at least 30 minutes to observe for any reactogenicity after immunization. Total follow-up is 90 days.

Blood specimens will be collected on Day 0 prior to vaccination, Day 21, Day 60, and day 90.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 18-49 years old
* Having Thai ID card or equivalent
* All hematology, biochemistry and urine analysis are within normal range or of no clinical significance (not higher than 1.5 time of normal value without any clinical finding from history and physical examination)
* Able to read and write and sign written informed consent form or assent form.

Exclusion Criteria:

* Known history of egg allergy
* Having had recently influenza infection confirmed as H1N1, H3N2, or Flu B within 3 months preceding enrolment to the trial
* Vaccination against influenza in the past 6 months preceding enrolment to the trial
* History of bronchial asthma, chronic lung diseases, chronic rhinitis
* History of immunodeficiency state
* History of immunosuppression < 6 months prior to immunization
* History of anaphylactic or other allergic reactions to influenza vaccine or any vaccine component or excipient (e.g. gentamicin or thimerosal)
* Acute infectious with fever > 38 degree Celsius and noninfectious diseases (within 72 hours) preceding enrollment in the trial
* The volunteers who have been taking immunoglobulin products or have had a blood transfusion during past 3 months before the beginning of the experiment
* Participation in other research study
* Pregnancy or plan to become pregnant for 60 days after enrollment or breast feeding
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled, or could interfere with the evaluation of the vaccine

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 340 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, Prof., Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 340 participants (40 in phase I and 300 in phase II) who met all inclusion criteria and not of the exclusion criteria were enrolled in the study.
Groups:
- Inactivated Influenza Vaccine Phase I; Inactivated Influenza Vaccine Phase II: A single dose of a seasonal trivalent inactivated split virion influenza vaccine [A/California/7/2009, reassortant virus NYMC X-181 (H1N1), A/Victoria/210/2009, reassortant virus NYMC X-187 (H3N2), and B/Brisbane/60/2008, reassortant virus NYMC BX-35 virus strains] 0.5 ml. was administered via the intramuscular route to the subjects at day 0 after blood collection for immunology assays.
- Placebo Phase I: A single dose of placebo (0.9% normal saline solution) 0.5 ml. was administered via the intramuscular route to the subjects at day 0 after blood collection for immunology assays.
- Placebo Phase II: A single dose of placebo (0.9% normal saline solution) was administered via the intramuscular route to the subjects at day 0 after blood collection for immunology assays.
Period: Overall Study
Arm/Group | Inactivated Influenza Vaccine Phase I | Placebo Phase I | Inactivated Influenza Vaccine Phase II | Placebo Phase II
Started | 20 | 20 | 200 | 100
Completed | 19 | 20 | 197 | 100
Not Completed | 1 | 0 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Phase II: A single dose of placebo (0.9% normal saline solution) 0.5 ml. was administered via the intramuscular route to the subjects at day 0 after blood collection for immunology assays.
- Total: Total of all reporting groups
Arm/Group | Inactivated Influenza Vaccine Phase I | Placebo Phase I | Inactivated Influenza Vaccine Phase II | Placebo Phase II | Total
Number analyzed (Participants) | 20 | 20 | 200 | 100 | 340
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 200 | 100 | 340
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Phase I and phase II was analyzed separately Phase I=40 (20 received vaccine, 20 received placebo).Phase II=300(ITT analysis). 200 received vaccine,100 received placebo).
  years | 32.25 (9.45) | 28.15 (6.72) | 32.28 (8.19) | 32.2 (7.96) | 31.22 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Phase I and phase II was analyzed separately. Numbers in phase I = 40, Phase II = 300 (Intent to treat analysis).
  Participants
    Female | 10 | 5 | 112 | 65 | 192
    Male | 10 | 15 | 88 | 35 | 148
Region of Enrollment [Count of Participants; unit: Participants] — Phase I: N=40 participants, Phase II: N = 300 participants
  Participants
    Thailand | 20 | 20 | 200 | 100 | 340

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: All Adverse Events during 90 days will be analysed in terms of percentage and relationship to study vaccine
Time Frame: 90 days
Population: All participants who receive at least one vaccination would be included in the safety population. The analysis will be conducted based on intent-to-treat (ITT) analysis. The population for the ITT analysis is defined as all individuals in the trial. The ITT analysis would include individuals who may not complete follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Inactivated Influenza Vaccine Phase I: Number of Participants With Adverse Events Phase I: AE/SAE Vaccine group (N=20)
- Placebo Phase I: Number of Participants With Adverse Events Phase I: AE/SAE Placebo group (N = 20)
- Inactivated Influenza Vaccine Phase II: Number of Participants With Adverse Events Phase II: AE/SAE Vaccine group (N=200)
- Placebo Phase II: Number of Participants With Adverse Events Phase II: AE/SAE placebo group (N=100)
Arm/Group | Inactivated Influenza Vaccine Phase I | Placebo Phase I | Inactivated Influenza Vaccine Phase II | Placebo Phase II
Number analyzed (Participants) | 20 | 20 | 200 | 100
Participants | 5 | 8 | 69 | 30

2. Secondary Outcome: Number (Percentage) of Participants With Achieving Seroconversions or Significant Increase in Antihemagglutinin Antibody Titer.
Description: Seroconversion is defined as a 4-fold rise in HAI titer in post-immunization serum relative to pre-immunization serum, or if pre-immunization serum had an undetectable titer (<1:10), attainment of a post-immunization titer of ≥1:40.
Time Frame: 90 days
Population: Seroconversion against the hemagglutinin antigens contained in the vaccine were assessed in all studied participants both phase I and phase II. The analysis was performed as intention-to-treat (ITT).
Measure: Count of Participants; unit: Participants
Arm/Group | Inactivated Influenza Vaccine Phase I | Placebo Phase I | Inactivated Influenza Vaccine Phase II | Placebo Phase II
Number analyzed (Participants) | 20 | 20 | 200 | 100
Participants
  A/H1N1 Day 21 | 17 | 0 | 176 | 0
  A/H1N1 Day 60 | 14 | 0 | 166 | 0
  A/H1N1 Day 90 | 13 | 0 | 163 | 1
  A/H3N2 day 21 | 9 | 1 | 107 | 0
  A/H3N2 Day 60 | 8 | 1 | 93 | 1
  A/H3N2 Day 90 | 7 | 1 | 92 | 2
  B/Brisbane/60/2008 Day 21 | 19 | 0 | 173 | 1
  B/Brisbane/60/2008 Day 60 | 19 | 2 | 153 | 1
  B/Brisbane/60/2008 Day 90 | 18 | 1 | 146 | 1

3. Secondary Outcome: Geometric Mean of Immune Response at Every Time of Assessment
Description: The analysis was performed only as intention-to-treat (ITT). The antibody titer values were transformed into log10 titers for calculation of the GMT at every time of assessment (Days 0,21, 60 and 90)
Time Frame: 90 days
Population: The antibody titer values were transformed into log10 titers for calculation of the GMT at every time of assessment (Days 0,21, 60 and 90) were assessed in all studied participants both phase I and phase II. The analysis was performed as intention-to-treat (ITT).
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Inactivated Influenza Vaccine Phase I | Placebo Phase I | Inactivated Influenza Vaccine Phase II | Placebo Phase II
Number analyzed (Participants) | 20 | 20 | 200 | 100
titer
  A/H1N1 Day 0 | 21.44 [11.12 to 41.33] | 24.62 [14.09 to 43.02] | 19.39 [16.40 to 22.92] | 20.14 [15.90 to 25.52]
  A/H1N1 Day 21 | 380.55 [246.97 to 586.38] | 24.62 [14.09 to 43.02] | 392.60 [337.59 to 456.59] | 20.00 [15.79 to 25.33]
  A/H1N1 Day 60 | 226.27 [149.51 to 342.45] | 24.62 [14.09 to 43.02] | 253.10 [218.31 to 293.42] | 20.00 [15.82 to 25.29]
  A/H1N1 Day 90 | 206.55 [133.78 to 318.90] | 24.62 [14.09 to 43.02] | 221.21 [189.48 to 258.25] | 20.85 [16.45 to 26.42]
  A/H3N2 Day 0 | 62.77 [40.53 to 97.21] | 64.98 [40.54 to 104.16] | 51.16 [43.43 to 60.27] | 44.38 [35.03 to 56.22]
  A/H3N2 Day 21 | 177.53 [128.84 to 244.61] | 72.10 [43.87 to 118.49] | 214.81 [183.77 to 251.09] | 43.17 [34.20 to 54.49]
  A/H3N2 Day 60 | 149.29 [109.06 to 204.35] | 72.10 [43.87 to 118.49] | 165.12 [143.17 to 190.43] | 43.17 [34.20 to 54.49]
  A/H3N2 Day 90 | 148.74 [111.03 to 199.26] | 69.64 [43.19 to 112.29] | 155.06 [135.47 to 177.48] | 45.00 [35.77 to 56.62]
  B/Brisbane/60/2008 Day 0 | 9.01 [6.54 to 12.42] | 14.14 [9.34 to 21.40] | 9.97 [8.72 to 11.39] | 9.20 [7.77 to 10.90]
  B/Brisbane/60/2008 Day 21 | 190.27 [110.26 to 328.35] | 13.66 [9.03 to 20.67] | 115.92 [97.60 to 137.66] | 9.40 [7.83 to 11.28]
  B/Brisbane/60/2008 Day 60 | 134.54 [79.60 to 227.43] | 16.82 [10.28 to 27.51] | 83.72 [70.39 to 99.58] | 9.33 [7.82 to 11.13]
  B/Brisbane/60/2008 Day 90 | 107.11 [61.16 to 187.58] | 15.69 [10.13 to 24.30] | 73.33 [61.15 to 87.94] | 9.40 [7.89 to 11.19]

4. Secondary Outcome: Geometric Mean of Immune Response Increase > 2.5 From Baseline of H1N1,H3N2 and B/Brisbane/60/2008 Antibody Titer
Description: The analysis was performed only as intention-to-treat (ITT). The antibody titer values were transformed into log10 titers for calculation of the GMT at every time of assessment (Days 0, 21, 60 and 90). Proportion of increased in GMT Titer > 2.5 at each time of assessment compared with baseline (Day 0) was reported both phase I and phase II
Time Frame: 90 days
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Inactivated Influenza Vaccine Phase I | Placebo Phase I | Inactivated Influenza Vaccine Phase II | Placebo Phase II
Number analyzed (Participants) | 20 | 20 | 200 | 100
titer
  A/H1N1 Day 21 | 17.75 [8.18 to 38.55] | 1.00 [1.00 to 1.00] | 20.25 [16.54 to 24.79] | 0.99 [0.97 to 1.02]
  A/H1N1 Day 60 | 10.56 [5.08 to 21.95] | 1.00 [1.00 to 1.00] | 13.06 [10.82 to 15.76] | 0.99 [0.97 to 1.02]
  A/H1N1 Day 90 | 9.26 [4.40 to 19.47] | 1.00 [1.00 to 1.00] | 11.45 [9.51 to 13.80] | 1.04 [0.96 to 1.11]
  A/H3N2 day 21 | 2.83 [1.70 to 4.71] | 1.11 [0.89 to 1.38] | 4.20 [3.47 to 5.07] | 0.97 [0.94 to 1.01]
  A/H3N2 Day 60 | 2.38 [1.52 to 3.71] | 1.11 [0.89 to 1.38] | 3.19 [2.71 to 3.75] | 0.97 [0.92 to 1.02]
  A/H3N2 Day 90 | 2.31 [1.43 to 3.74] | 1.07 [0.85 to 1.35] | 3.03 [2.60 to 3.53] | 1.01 [0.96 to 1.08]
  B/Brisbane/60/2008 Day 21 | 21.11 [12.97 to 34.35] | 0.97 [0.90 to 1.04] | 11.63 [9.68 to 13.98] | 1.02 [0.95 to 1.10]
  B/Brisbane/60/2008 Day 60 | 14.93 [9.23 to 24.15] | 1.19 [0.92 to 1.53] | 8.40 [6.99 to 10.10] | 1.01 [0.95 to 1.09]
  B/Brisbane/60/2008 Day 90 | 12.85 [8.23 to 20.08] | 1.11 [0.92 to 1.34] | 7.33 [6.08 to 8.84] | 1.02 [0.95 to 1.10]

ADVERSE EVENTS:
Time Frame: 90 days
Groups:
- Inactivated Influenza Vaccine Phase I: Serious Adverse Event Phase I vaccine group N= 20
- Placebo Phase I: Serious Adverse Event Phase I placebo group N= 20
- Inactivated Influenza Vaccine Phase II: Serious Adverse Event Phase I vaccine group N= 200
- Placebo Phase II: Serious Adverse Event Phase I placebo group N= 100
Arm/Group | Inactivated Influenza Vaccine Phase I | Placebo Phase I | Inactivated Influenza Vaccine Phase II | Placebo Phase II
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/200 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/200 | 0/100
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/200 | 0/100

LIMITATIONS AND CAVEATS:
No limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No